CLINICAL TRIAL: NCT01328613
Title: A Prospective Study of Postpartum Depression in Women With Major Depression
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908320; 08-AG-N320
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2014-09-29

CONDITIONS: Postpartum Depression
Keywords: BDNF; Homeosis; Women; Childbirth; Major Depressive Disorder
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Postpartum depression (PPD) is a serious syndrome that resembles a major depressive episode and occurs in 10% to 20% of all mothers in the year following delivery. Women with histories of major depressive disorder (MDD) are at an increased risk for PPD and recurrent PPD with subsequent pregnancies. One possible genetic vulnerability to depression and PPD in particular is the BDNF gene. BDNF is a protein that affects the growth and development of brain cells, including those that help to regulate mood. BDNF levels have been shown to be significantly lower in individuals with depression, including women. Researchers are interested in studying BDNF levels and hormones such as estrogen in pregnant women who have MDD and are at risk for developing PPD.

Objectives:

- To study connections between the BDNF protein and hormonal levels in pregnant women who are at risk for developing postpartum depression.

Eligibility:

- Women who are currently pregnant and have a history of major depressive disorder, and either are taking a selective serotonin reuptake inhibitor (SSRI) or are not taking an antidepressant.

Design:

* This study involves six visits over the course of 12 months, during the first, second, and third trimesters (if possible) as well as 1 week, 1 month, and 3 months postpartum. Women will be allowed to participate at any point during pregnancy, but researchers are most interested in recruiting women who are in the first trimester.
* Participants will be screened with a physical examination and medical history, blood samples, and questionnaires about their history of depressive episodes.
* At each visit, participants will complete a number of questionnaires on depression symptoms, such as sleep disturbance and stress levels. Participants will also provide blood samples for hormone and other testing.
* Participants who become depressed during the study will be referred to a treating psychiatrist or other professional for appropriate care and treatment.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a serious syndrome which resembles a major depressive episode and occurs in 10-20% of all mothers in the year following delivery. The etiology of PPD involves psychological factors, environmental factors such as stress and sleep deprivation, biological factors including hormonal changes, and social factors. Women with histories of major depression (MDD) are at an increased risk for PPD and recurrent PPD with subsequent pregnancies. No consistent hormonal abnormalities have been found in women with PPD and, instead, they may be sensitive to the normal changes in hormone levels during the postpartum time. One possible genetic vulnerability to depression, and in particular PPD, is the brain-derived neurotrophic factor (BDNF) gene. BDNF is an important member of the neurotrophin family and is known to affect neuronal outgrowth, differentiation, synaptic connectivity and neuronal repair for a broad range of neuronal cell types including serotonergic neurons. In humans, serum BDNF levels have been shown to be significantly lower in patients with depression, including women . Interestingly, estrogen has been shown to upregulate the expression of the BDNF gene in animals, suggesting that BDNF could be a critical link for women who have hormonally related depressive symptoms. In addition, serotonin-selective reuptake inhibitors (SSRI) used to treat depression are known to upregulate the expression of BDNF in the brain. Interestingly, links between depression, perturbed energy metabolism and BDNF signaling have recently been elucidated. In the present study, NIA investigators will measure levels of BDNF and reproductive and energy-regulating hormones in serum samples from subjects enrolled in Dr. Jennifer Payne s study of PPD.

All subjects in this study will be enrolled, evaluated and serum samples collected by Dr. Payne and her staff at Johns Hopkins University School of Medicine under Dr. Payne s already Johns Hopkins approved IRB protocol NA_0008149.

NIA Role:

Coded serum samples will then be sent to Dr. Mattson at the NIA facility. Data obtained in the analysis of serum samples will be sent to Dr. Payne and maintained in her database, and analyzed to elucidate relations between levels of serum markers and clinical and genetic data acquired by Dr. Payne.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women who are currently pregnant and who have a history of MDD.

In order to minimize heterogeneity in the sample, all women must be currently taking a serotonin reuptake inhibitor (SSRI) antidepressant medication or not taking antidepressants.

We will attempt to recruit approximately 50% in each category (SSRI versus no medications). If a woman becomes depressed during the study she will be referred to her treating psychiatrist or given appropriate clinical care. We will continue to follow women for the specified time course even if she placed on an (any) antidepressant medication during the course of the study.

EXCLUSION CRITERIA:

Diagnosis of bipolar disorder

Current active suicidal ideation or medical instability

Active substance abuse or dependence during the last 90 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-11-09; Study Completion 2014-09-29

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Mattson, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Campbell SB, Cohn JF. Prevalence and correlates of postpartum depression in first-time mothers. J Abnorm Psychol. 1991 Nov;100(4):594-9. doi: 10.1037//0021-843x.100.4.594. PMID 1757673
- [Background] Hunt N, Silverstone T. Does puerperal illness distinguish a subgroup of bipolar patients? J Affect Disord. 1995 May 17;34(2):101-7. doi: 10.1016/0165-0327(95)00006-9. PMID 7665801
- [Background] Kumar R, Robson KM. A prospective study of emotional disorders in childbearing women. Br J Psychiatry. 1984 Jan;144:35-47. doi: 10.1192/bjp.144.1.35. PMID 6692075